CLINICAL TRIAL: NCT04911582
Title: Does the Bioactive Substance in Coffee, Cafestol, Have Preventive Properties on Type-2-diabetes? Acute and Longer-term Metabolic Effects of Cafestol. (Acute Substudy)
Brief Title: Does the Bioactive Substance in Coffee, Cafestol, Have Preventive Properties on Type-2-diabetes? (Acute Substudy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cafestol.acute.waist
Record Dates: First submitted 2021-05-27; First posted 2021-06-03 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-05

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — cafestol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cafestol 6 mg (Active Comparator): 6 mg cafestol
  Interventions: Dietary Supplement: Cafestol 6 mg
- Cafestol 12 mg (Active Comparator): 12 mg cafestol
  Interventions: Dietary Supplement: Cafestol 12 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cafestol 12 mg — Capsule with 12 mg cafestol
  Arms: Cafestol 12 mg
Dietary Supplement: Placebo — Placebo capsule without cafestol
  Arms: Placebo
Dietary Supplement: Cafestol 6 mg — Capsule with 6 mg cafestol
  Arms: Cafestol 6 mg

SUMMARY:
Acute, double-blinded, randomized, cross-over cafestol intervention study with fifteen participants with a large waist circumference participating in three OGTTs.

DETAILED DESCRIPTION:
The study is a acute, double-blinded, randomized, controlled intervention in 15 subjects with abdominal obesity at high risk of developing T2D. Initially, a blood sample is obtained (t=-15 min) and at time point 0, the participants will ingest a capsule containing either 6 or 12mg cafestol or placebo. Immediately hereafter an OGTT commences with ingestion of a 75 g glucose solution. In the following 2 hours blood samples are collected at time points 15, 30, 60, 90, 120 and 180 min. The samples will be used for determination of plasma glucose, insulin and cafestol, as well as GLP-1 and GIP. After a one-week washout period, the subject will undergo the same set-up again, however now with the different dosage of cafestol or placebo. The process is repeated for three weeks until every subject has undergone both interventions and the placebo.

ELIGIBILITY:
Inclusion Criteria:

25 < BMI < 40 kg/m2 Waist circumference > 102 cm (men) / 88 cm (women)

Exclusion Criteria:

* Type 2 diabetes (HbA1c > 48 mmol/mol) or in treatment with antidiabetic drugs
* Pregnancy
* Planned pregnancy
* Breastfeeding
* Significant comorbidity expected to unable the subject from completing visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve for glucose | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for glucose during OGTT after ingestion of cafestol or placebo capsule (mmol/L)

SECONDARY OUTCOMES:
Area under the curve for insulin-response | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for insulin response during OGTT after ingestion of cafestol or placebo capsule (pmol/L)
Area under the curve for cafestol | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for cafestol during OGTT after ingestion of cafestol or placebo capsule
Area under the curve for GLP-1 (glucagon-like peptide-1) | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for GLP-1 (glucagon-like peptide-1) during OGTT after ingestion of cafestol or placebo capsule (pmol/L)
Area under the curve for GIP (Glucose-dependent insulinotropic polypeptide) | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for GIP (Glucose-dependent insulinotropic polypeptide) during OGTT after ingestion of cafestol or placebo capsule (pmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided